CLINICAL TRIAL: NCT02212431
Title: An Open Label Investigation of the Tolerability and Pharmacokinetics of Oral Cysteamine in Adults With Cystic Fibrosis.
Brief Title: First Study of Oral Cysteamine in Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Cystic Fibrosis Trust (Other); NHS Grampian (Other Government); University of Huddersfield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 3/001/14; 2014-000284-40 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Cysteamine; Pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cysteamine (Experimental): Dosing will be in accordance with licensed use of cysteamine for cystinosis, i.e. 450mg qds.
  Dose will be escalated:
  450mg od for one week 450mg bd for one week 450mg tds for one week 450mg qds for two weeks
  Interventions: Drug: Cysteamine

INTERVENTIONS:
Drug: Cysteamine — Dose will be increased weekly from 450mg od to 450mg bd, to 450mg tds to 450mg qds, will remain on highest dose for 2 weeks
  Other Names: Cystagon 150mg capsules

SUMMARY:
The morbidity and mortality associated with Cystic Fibrosis (CF) are the result of chronic suppurative lung disease. The aggressive use of antibiotics is one of the mainstays of treatment in CF, however, the problems of multiple drug resistance and adverse reactions are major clinical issues.

Cysteamine is a licensed drug used in the treatment of cystinosis. In vitro work suggests that cysteamine has properties of potential benefit in CF. Cysteamine is a potent mucolytic, it disrupts biofilms, it is antimicrobial, and synergises with other antibiotic agents. CF is characterised by malabsorption and it is not known whether cysteamine is absorbed in CF, furthermore it is not known if cysteamine enters the bronchial secretions. It is not possible to assume that the pharmacokinetics of cysteamine in patients with CF are the same as those reported for cystinosis.

Objectives: to characterise the pharmacokinetic profile of cysteamine in people with CF, to ascertain whether cysteamine enters the bronchial secretions and the tolerability of cysteamine by patients with CF.

Method: a single centre, single group open label investigation of the tolerability and pharmacokinetics of oral cysteamine (Cystagon) when administered to patients with Cystic Fibrosis at the dose licensed for use in cystinosis.

Setting: adult CF clinic, Aberdeen Royal Infirmary.

Target population: 12 patients aged ≥18years with CF associated lung disease who are clinically stable.

Intervention: Oral cysteamine (Cystagon) will be increased from 450mg od to 450mg qds over three weeks, they will remain on 450mg qds for two weeks.

Assessment: face to face health outcome assessments will be carried out for all participants at recruitment/baseline, 1, 2, 3, and 5 and 6 weeks. Serial blood cysteamine levels will be measured in the first 24 hours after the first dose. Sputum cysteamine will be quantified after two weeks of full dose cysteamine 450mg qds. Disease specific health status (CFQ-R) will be assessed at baseline and after two weeks of full dose. At each assessment, lung function (FEV1, FVC), adverse reactions and serious adverse events will be ascertained. Blood samples will be taken for measurement of haematological and biochemical parameters. Sputum samples at each assessment will be analysed for microbial load and spinnbarkeit.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is the commonest fatal inherited disease in Caucasian populations of European origin. The morbidity and mortality associated with CF are the result of chronic suppurative lung disease. The lungs of people with CF are chronically infected with bacteria that cause chronic infection and acute periods of worsening infection known as exacerbations. Many of the bacteria that infect patients with CF are intrinsically resistant to many antibiotics and bacterial antibiotic resistance is increasing, in addition many of the pathogenic bacteria grow in biofilms that contributes to antibiotic resistance. The aggressive use of antibiotics to suppress chronic infection and to treat acute exacerbations is one of the mainstays of treatment in CF that has contributed to the increased survival of CF patients. However, the problems of multiple drug resistance and adverse reactions are major clinical issues. This has led to calls for research into new antibiotics and new antibiotic strategies to target the biofilm and to increase the effectiveness of currently available antibiotics.

Cysteamine is a licensed drug used in the treatment of cystinosis for more than 20 years. Laboratory based work suggests that cysteamine may be a beneficial adjunct to conventional antibiotic treatment in CF. Cysteamine is a potent mucolytic, it disrupts biofilms, it is antimicrobial, and synergises with other antibiotic agents, broadening their spectrum of activity, delivers a post-antimicrobial effect and reverses antibiotic resistance (even in multi-drug resistant bacteria). Although the pharmacokinetic characteristics of cysteamine are well established in people with cystinosis, there are no such data for cysteamine in CF. CF is characterised by malabsorption and it is not known whether cysteamine is absorbed in CF, furthermore it is not known if cysteamine enters the bronchial secretions. It is not possible to assume that the pharmacokinetics of cysteamine in patients with CF are the same as those reported for cystinosis.

Hypothesis: Oral cysteamine will be absorbed into the vascular space and bronchial secretions after administration to people with Cystic Fibrosis.

Objectives: to characterise the pharmacokinetic profile of cysteamine in people with CF, to ascertain whether cysteamine enters the bronchial secretions and the tolerability of cysteamine by patients with CF.

Method: a single centre, single group open label investigation of the tolerability and pharmacokinetics of oral cysteamine (Cystagon) when administered to patients with Cystic Fibrosis at the dose licensed for use in cystinosis.

Setting: adult CF clinic, Aberdeen Royal Infirmary.

Target population: 12 patients aged ≥18years with CF associated lung disease who are clinically stable.

Intervention: as recommended for cystinosis, patients will be maintained on their normal CF medication. Oral cysteamine (Cystagon) will be increased from 450mg od to 450mg qds over three weeks, they will remain on 450mg qds for two weeks.

Assessment: face to face health outcome assessments will be carried out for all participants at recruitment/baseline, 1, 2, 3, and 5 and 6 weeks. Serial blood cysteamine levels will be measured in the first 24 hours after the first dose. Sputum cysteamine will be quantified after two weeks of full dose cysteamine 450mg qds. Disease specific health status (CFQ-R) will be assessed at baseline and after two weeks of full dose. At each assessment, lung function (FEV1, FVC), adverse reactions and serious adverse events will be ascertained. Blood samples will be taken for measurement of haematological and biochemical parameters that are recognised, but rare side effects of cysteamine. Sputum samples at each assessment will be analysed microbiologically (quantitative, antibiotic sensitivity and rheology) to assess effects of cysteamine on sputum microbiology, sputum collected prior to first dosing will be used to develop a laboratory based method to quantify cysteamine in sputum.

ELIGIBILITY:
Inclusion Criteria:

* CF related suppurative lung disease who expectorate sputum,
* Clinically stable for >4 weeks,
* Aged ≥18 years,
* Weight >50kg,
* Female participants of child bearing potential should be using a reliable form of contraception.

Exclusion Criteria:

* Hypersensitivity to the active substance, any form of cysteamine, or to any of the excipients.
* Hypersensitivity to penicillamine.
* Lung, liver transplant, on active transplant list.
* For women, current pregnancy or breast-feeding, or planned pregnancy during the study.
* Any other significant disease/disorder which, in the investigator's opinion, either puts the patient at risk because of study participation or may influence the results of the study or the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Elimination rate constant [k] | 24 hours
  Blood cysteamine prior to the initial dose on day 1 and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours post-dose

SECONDARY OUTCOMES:
Concentration of cysteamine in sputum at week 5 | 3 hours after final dose

OTHER OUTCOMES:
Change in weight from baseline at week 5 | 5 weeks
Number of Participants with Serious and Non-Serious Adverse Events | 6 weeks
Change in FEV1, FVC from baseline at week 5 | 5 weeks
Change in disease related health status from baseline at week 5 measured by CFQ-R | 5 weeks
Change in haematological and biochemical indices from baseline at week 5 | 5 weeks
change in sputum microbiology from baseline at week 5 | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graham Devereux, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom